CLINICAL TRIAL: NCT00253383
Title: Improving Palliative Care for Patients With Cancer
Brief Title: Early Intervention vs. Standard Palliative Care in Improving End-of-Life Care in Advanced Cancer Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Dartmouth-Hitchcock Medical Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: CDR0000452966; R01CA101704 (NIH); P30CA023108 (NIH); DMS-0226; DMS-CPHS-16004
Record Dates: First submitted 2005-11-11; First posted 2005-11-15 (Estimated); Last update posted 2014-12-19 (Estimated); Status verified 2014-12

CONDITIONS: Cancer
Keywords: transitional care planning; stage IIIB non-small cell lung cancer; stage IV non-small cell lung cancer; extensive stage small cell lung cancer; stage IV breast cancer; recurrent breast cancer; male breast cancer; stage IIIB anal cancer; stage IV anal cancer; carcinoma of the appendix; stage III colon cancer; stage IV colon cancer; stage III rectal cancer; stage IV rectal cancer; stage III esophageal cancer; stage IV esophageal cancer; unresectable extrahepatic bile duct cancer; unresectable gallbladder cancer; stage III gastric cancer; stage IV gastric cancer; metastatic gastrointestinal carcinoid tumor; regional gastrointestinal carcinoid tumor; gastrointestinal stromal tumor; advanced adult primary liver cancer; localized unresectable adult primary liver cancer; stage III pancreatic cancer; recurrent small intestine cancer; small intestine adenocarcinoma; small intestine leiomyosarcoma; small intestine lymphoma; stage IV bladder cancer; stage IV renal cell cancer; clear cell sarcoma of the kidney; peripheral primitive neuroectodermal tumor of the kidney; rhabdoid tumor of the kidney; metastatic transitional cell cancer of the renal pelvis and ureter; anterior urethral cancer; posterior urethral cancer; urethral cancer associated with invasive bladder cancer; stage IV penile cancer; stage IV prostate cancer; stage III malignant testicular germ cell tumor; stage IV endometrial carcinoma; fallopian tube cancer; ovarian sarcoma; ovarian stromal cancer; stage IV pancreatic cancer
MeSH Terms: conditions — Neoplasms; Carcinoma, Non-Small-Cell Lung; Breast Neoplasms; Breast Neoplasms, Male; Anus Neoplasms; Appendiceal Neoplasms; Colonic Neoplasms; Rectal Neoplasms; Esophageal Neoplasms; Stomach Neoplasms; Gastrointestinal Stromal Tumors; Pancreatic Neoplasms; Urinary Bladder Neoplasms; Carcinoma, Renal Cell; Penile Neoplasms; Prostatic Neoplasms; Testicular Neoplasms; Endometrial Neoplasms; Fallopian Tube Neoplasms | interventions — Counseling; Early Intervention, Educational; Psychiatric Rehabilitation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- ENABLE (concurrent palliative care) (Experimental): telephone based ENABLE educational intervention
  Interventions: Other: counseling intervention; Other: educational intervention; Procedure: psychosocial assessment and care; Procedure: quality-of-life assessment
- Usual Care (Active Comparator): Supportive and palliative usual care services at DHMC, Behavioral
  Interventions: Other: counseling intervention; Procedure: psychosocial assessment and care; Procedure: quality-of-life assessment

INTERVENTIONS:
Other: counseling intervention
Other: educational intervention
  Arms: ENABLE (concurrent palliative care)
Procedure: psychosocial assessment and care
Procedure: quality-of-life assessment

SUMMARY:
RATIONALE: Palliative care may help patients with advanced cancer live more comfortably.

PURPOSE: This randomized clinical trial is studying an early intervention palliative care program to see how well it works compared to a standard care program in improving end-of-life care in patients with advanced lung , gastrointestinal, genitourinary, or breast cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the efficacy of an early intervention palliative care program comprising a phone-based nurse educator and shared medical appointments in improving end-of-life care of patients with advanced lung, gastrointestinal, genitourinary, or breast cancer.
* Compare symptom management, quality of life, and the match between preference of care and the care received in patients treated with an early intervention palliative care program vs a standard care program.
* Compare health care utilization by patients treated with these interventions.

OUTLINE: This is a randomized, multicenter study. Patients are stratified according to cancer diagnosis (lung vs breast vs gastrointestinal vs genitourinary) and participating center. Patients are randomized to 1 of 2 intervention arms.

* Arm I (early-intervention palliative care program): Patients complete the Medical Care Questionnaire and receive a computer-generated prescription letter that outlines the problems they have identified; the patient's physician also receives a copy of the letter. Patients receive a series of phone calls weekly for 4 weeks and then at least monthly from a nurse educator. The phone calls address 3 major areas: coordination of palliative care options in the cancer center and the patient's community, including referrals for psychological or spiritual counseling, social work consultation, financial guidance, home health, palliative care or hospice services, and bereavement counseling for the family; problem-solving therapy, focusing on the identification of problems, definition of achievable goals, a plan for reaching those goals, and evaluation of success; and tailored psycho-educational modules from "Charting Your Course", covering end-of-life topics such as symptom management, advanced care planning, communication with the health care team and family members, spirituality, and nutrition. Patients also receive information regarding the purpose and time/location of symptom management, shared medical appointments (SMAs), which they can attend in person or call in to participate via speaker phone. SMAs are 1.5-hour monthly sessions conducted by a physician and a nurse practitioner that can accommodate 10-12 patients and their caregivers. The sessions include a welcome/social period, a question and answer/peer discussion, an interactive educational session, and an opportunity for one-on-one nurse practitioner appointments with a focus on a brief review of the patients' medical treatment plans.
* Arm II (standard palliative care program): Patients receive standard palliative care from their physician/nurse practitioner team and have access to the palliative care nurse at the discretion of the treating physician.

Patients complete Functional Assessment of Chronic Illness Therapy-Palliative Care at baseline and every 3 months thereafter. Patients and caregivers complete surveys measuring their perception of the quality of the patient's cancer care at baseline and at 1 month.

A caregiver or family member completes the After-Death Bereaved Family Member Interview to evaluate the adequacy of patient care at 3 months post-patient death.

PROJECTED ACCRUAL: A total of 450 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Diagnosis of 1 of the following advanced cancers:

  * Stage IIIB or IV non-small cell lung cancer
  * Extensive stage small cell lung cancer
  * Stage IV breast cancer

    * Poor prognostic indicators (conferring likelihood of ≤ 2 years survival), including, but not limited to, any of the following:

      * Visceral crisis
      * Lung or liver metastasis
      * Estrogen receptor-negative disease
      * HER2/neu-positive disease
      * Progressive or recurrent disease during or within 2 years of first treatment
  * Unresectable stage III or stage IV gastrointestinal cancers
  * Stage IV genitourinary cancers

    * Prostate cancer must be hormone refractory
* Hormone receptor status:

  * Not specified

PATIENT CHARACTERISTICS:

Sex

* Not specified

Menopausal status

* Not specified

Performance status

* Not specified

Life expectancy

* Not specified

Hematopoietic

* Not specified

Hepatic

* Not specified

Renal

* Not specified

Other

* No dementia or significant confusion (i.e., Mini Mental Exam score < 25)
* No Axis I psychiatric disorders (DSM-IV), including any of the following:

  * Schizophrenia
  * Bipolar disorder
  * Active substance use disorder

PRIOR CONCURRENT THERAPY:

Endocrine therapy

* See Disease Characteristics

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 329 (Actual)
Dates: Start 2003-01; Primary Completion 2013-09 (Actual); Study Completion 2013-09 (Actual)

PRIMARY OUTCOMES:
Quality of life as measured by Functional Assessment of Cancer Therapy-Palliative care version (FACT-Pal) at baseline, one month, and every three months thereafter | Baseline, one month, every three months
Symptom management as measured by Edmunton Symptom Assessment Scale at baseline, one month, and every three months thereafter | Baseline, one month, every three months
Health care utilization by a chart review of days in hospital, ICU, ER visits at baseline, one month, and every three months thereafter | Baseline, one month, every three months
Correlate preferences for care and care received as measured by After Death Bereaved Family Member Interview with a family member of the deceased | Baseline, one month, every three months

SECONDARY OUTCOMES:
Depression as measured by Center for Epidemiological Studies-Depression (CES-D) at baseline, one month, and every three months thereafter | Baseline, one month, every three months
Problem solving skills as measured by Social Problem-Solving Skills Inventory-revised at baseline and one month | Baseline, one month, every three months
Caregiver burden as measured by Montgomery-Borgatta Caregiver Burden Scale at baseline, one month, and every three months thereafter (given to caregivers of patients) | Baseline, one month, every three months

CONTACTS AND LOCATIONS:
Overall Officials: Marie A Bakitas, PhD, Principal Investigator — Norris Cotton Cancer Center
Locations (2):
- United States (2):
  - Norris Cotton Cancer Center at Dartmouth-Hitchcock Medical Center, Lebanon, New Hampshire
  - Veterans Affairs Medical Center - White River Junction, White River Junction, Vermont

REFERENCES:
- [Result] Bakitas M, Lyons KD, Hegel MT, Balan S, Brokaw FC, Seville J, Hull JG, Li Z, Tosteson TD, Byock IR, Ahles TA. Effects of a palliative care intervention on clinical outcomes in patients with advanced cancer: the Project ENABLE II randomized controlled trial. JAMA. 2009 Aug 19;302(7):741-9. doi: 10.1001/jama.2009.1198. PMID 19690306
- [Derived] Corn BW, Feldman DB, Hull JG, O'Rourke MA, Bakitas MA. Dispositional hope as a potential outcome parameter among patients with advanced malignancy: An analysis of the ENABLE database. Cancer. 2022 Jan 15;128(2):401-409. doi: 10.1002/cncr.33907. Epub 2021 Oct 6. PMID 34613617
- [Derived] Prescott AT, Hull JG, Dionne-Odom JN, Tosteson TD, Lyons KD, Li Z, Li Z, Dragnev KH, Hegel MT, Steinhauser KE, Ahles TA, Bakitas MA. The role of a palliative care intervention in moderating the relationship between depression and survival among individuals with advanced cancer. Health Psychol. 2017 Dec;36(12):1140-1146. doi: 10.1037/hea0000544. Epub 2017 Oct 19. PMID 29048177